CLINICAL TRIAL: NCT04968730
Title: Establishment and Application of Early Postoperative Activity Plan for Patients After Hemi-laminectomy for Lumbar Spinal Tumor Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-0116
Record Dates: First submitted 2021-06-01; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-05

CONDITIONS: Tumor of Spinal Cord
Keywords: early rehabilitation training
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Intervention Model Description: The routine group was given routine nursing, and the control group was given early rehabilitation nursing
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group A (Placebo Comparator): routine nursing after operation
  Interventions: Other: Postoperative rehabilitation nursing
- intervention group B (Experimental): Nursing care after operation with stage intervention
  Interventions: Other: Postoperative rehabilitation nursing

INTERVENTIONS:
Other: Postoperative rehabilitation nursing — Make postoperative rehabilitation plan according to nursing experience for group A Develop rehabilitation process according to the activity plan for group B

SUMMARY:
Objective to construct the related early activity program for patients with lumbar intraspinal tumor after hemilaminectomy, and evaluate the postoperative limb function exercise according to the content of the program. In order to improve the self-care ability and quality of life of patients, reduce postoperative complications, shorten the average length of stay, reduce hospitalization expenses and improve patient satisfaction.

Objective to evaluate the efficacy and safety of establishing early activity program after hemilaminectomy for patients with lumbar intraspinal tumors

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary benign intraspinal tumors at the level of L1-L5 who underwent semi laminectomy;
2. The age of the patients ranged from 14 to 80 years old;
3. The GCS score was 15 points, and the lower limb muscle strength was more than or equal to grade 3 before operation; The patients agreed to the operation and were willing to accept and cooperate with the concept of early rehabilitation nursing and related measures;

Exclusion Criteria:

1. patients with rapid development of disease, difficult to exclude malignant tumors, and non neoplastic lesions in spine or spinal canal;
2. Have a history of severe hypertension, heart disease or other mental illness;
3. Patients with major organ damage or coagulation dysfunction;
4. The patients and their family members had poor communication and compliance;
5. There are factors that may progress or worsen the patient's condition (such as uncontrolled infection, severe respiratory disease, pulmonary infection, etc.);

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient rehabilitation and leave hospital | up to two years
  The whole clinical courses were strictly controlled in quality so as to compare the average length of stay (days) in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Wangping Neurosurgical, Hangzhou, China